CLINICAL TRIAL: NCT06012851
Title: Personalizing Behavioral Parent Training: Improving Reach and Outcomes for Families of Children With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Mobile Behavioral Parent Training for Childhood ADHD: A Micro-randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1R34MH128513-01 (NIH)
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: All participants receive access to a beta version of the mobile behavioral parent training application. Each participant is randomized multiple times per day (about 4-6 times per day) to received either no push notification (50% chance) or a push notification providing parenting feedback or a suggestion to use a parenting strategy (50% chance).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobile BPT with in-the-moment feedback (Experimental): Participants will be randomized multiple times per day to receive a push notification that provides feedback about parenting.
  Interventions: Behavioral: Mobile behavioral parent training (mBPT); Behavioral: In the moment feedback
- Mobile BPT with in-the-moment suggestions (Experimental): Participants will be randomized multiple times per day to receive a push notification that provides a suggestion for a parenting behavior.
  Interventions: Behavioral: Mobile behavioral parent training (mBPT); Behavioral: In the moment suggestions
- Mobile BPT only (Other): Participants will be randomized multiple times per day to receive no push notification.
  Interventions: Behavioral: Mobile behavioral parent training (mBPT)

INTERVENTIONS:
Behavioral: Mobile behavioral parent training (mBPT) — The mobile phone application includes behavioral parent training content (for example, praise, effective commands, reward systems) delivered in videos, examples, and quizzes that parents/caregivers access.
Behavioral: In the moment feedback — In-the-moment feedback will include parenting feedback.
  Arms: Mobile BPT with in-the-moment feedback
Behavioral: In the moment suggestions — In-the-moment feedback will include suggestions for parenting strategies.
  Arms: Mobile BPT with in-the-moment suggestions

SUMMARY:
The goal of the study is to develop and refine a personalized behavioral parent training intervention for caregivers of children with attention deficit hyperactivity disorder (ADHD). The behavioral intervention will teach positive parenting through videos and quizzes that caregivers can access through a smartphone application. The program also gives parents and caregivers in-the-moment feedback their use of parenting strategies. The current study, a micro-randomized trial, aims to see whether the in-the-moment feedback given to parents (a push notification on their smartphone) changes parenting behavior right after the feedback. Micro-randomized means that parents are randomly assigned repeatedly, in this study multiple times per day, to receive or not receive parenting feedback or suggestions on their smartphones.

The main questions to answer are:

Is parenting feedback provided by a smartphone application acceptable to caregivers? When parents receive the feedback, do they use more positive parenting skills in the next few minutes compared to when they do not receive the feedback? Is the phone application usable and acceptable to parents and caregivers of children with attention deficit hyperactivity disorder?

ELIGIBILITY:
Inclusion Criteria:

* Currently meets Diagnostic Statistical Manual 5 diagnostic criteria for ADHD
* Ages 7 -12
* Has parent-reported impairment in homework performance defined as a score of 3 or greater on an Impairment Rating Scale measure (Fabiano et al., 2006) of homework performance
* Has at least one parent or primary caregiver who is willing to participate and is able to access the intervention at home via smartphone.

Exclusion Criteria:

* N/A

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Passive Audio Data-Positive Sentiment Analysis | Through study completion, average of 5 weeks
  Parent and child interaction behavior- proportion of recorded interaction that is labeled positive via sentiment analysis algorithm. This will be assessed during scheduled, daily audio recordings. Specifically, we will assess sentiment after the randomization of prompt delivery and prior to the next randomization.
Passive Audio Data-Negative Sentiment Analysis | Throughout study completion, average of 5 weeks
  Parent and child interaction behavior- proportion of recorded interaction that is labeled negative via sentiment analysis algorithm. This will be assessed during scheduled, daily audio recordings. Specifically, we will assess sentiment after the randomization of prompt delivery and prior to the next randomization.

SECONDARY OUTCOMES:
Intervention Engagement | Through study completion, average of 5 weeks
  Number of mobile BPT sessions completed divided by the total number of sessions available.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Children and Families of Western New York, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT06012851/ICF_000.pdf